CLINICAL TRIAL: NCT01207232
Title: The Effect of a Planning Prompt on Seasonal Influenza Vaccination Rates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Harvard University (Other); Yale University (Other); Stanford University (Other)
Responsible Party: Professor Katherine L. Milkman, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 810589-1
Record Dates: First submitted 2010-09-20; First posted 2010-09-22 (Estimated); Last update posted 2010-09-22 (Estimated); Status verified 2010-09

CONDITIONS: Seasonal Influenza
Keywords: seasonal influenza; behavioral economics; implementation intentions; planning prompt; nudge

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Time Plan Condition (Experimental): A basic reminder mailing prompted each subject to write down a planned date and time for getting their flu shot.
  Interventions: Behavioral: Planning Prompt
- Date Plan Condition (Experimental): A basic reminder mailing prompted each subject to write down a planned date for getting their flu shot.
  Interventions: Behavioral: Planning Prompt
- Control Condition (Active Comparator): A basic reminder mailing prompted each subject to receive a flu shot.
  Interventions: Behavioral: Control Condition

INTERVENTIONS:
Behavioral: Planning Prompt — A prompt to write down a planned date (or date and time) for getting a flu shot
  Arms: Date Plan Condition; Time Plan Condition
Behavioral: Control Condition — A basic reminder mailing prompted each subject to get their flu shot.
  Arms: Control Condition

SUMMARY:
The investigators conducted a 3-arm randomized controlled trial to test whether a low-cost planning intervention could increase influence vaccination rates.

DETAILED DESCRIPTION:
Seasonal influenza causes 20,000 hospitalizations and 36,000 deaths in the U.S. each year. Past psychology research has demonstrated that prompting people to form an implementation plan of the form, "When situation x arises, I will implement response y," increases attainment of desired goals because the desired behavior is linked to a concrete future moment. This type of planning prompt is a "nudge" in the direction of desired behavior that can be implemented at minimal expense and does not restrict individual autonomy. We conducted a 3-arm randomized controlled trial to test whether a low-cost planning intervention could increase influence vaccination rates. We show that planning prompts can be successfully applied to improve health behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Vaccine indications according to fall 2009 CDC criteria (age >= 50 or chronic disease
* Employee at partner corporation that implemented the study

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3272 (Actual)
Dates: Start 2009-10; Primary Completion 2009-11 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Receipt of 2009 Seasonal Influenza Vaccination | up to 30 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Katherine L Milkman, Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States